CLINICAL TRIAL: NCT02446301
Title: A Bioavailability Study of Sebacoyl Dinalbuphine Ester IM Injection vs. Bain®. Nalbuphine HCl IM Injection, in Healthy Volunteers
Brief Title: A Bioavailability Study of Sebacoyl Dinalbuphine Ester IM Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LT1001-103
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Pain; Analgesia Disorder
Keywords: Nalbuphine; SDE; dinalbuphine; SDN; pain; LT1001
MeSH Terms: conditions — Pain | interventions — Nalbuphine; sebacoyl dinalbuphine ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period I (reference drug) (Experimental): Before administration of investigational products, subjects should be fasted for 10 hours. On the dosing day, subjects will be confined after administration and won't be discharged until after completion of sample collections for 24 hours following dosing in Period I (Bain® IM injection).
  Interventions: Drug: Bain®
- Period II (Test drug) (Experimental): Subjects will be back to the clinical site to join Period II (SDE IM injection) and will be discharged after completion for sample collections for 24 hours post drug administration.
  Interventions: Drug: SDE

INTERVENTIONS:
Drug: Bain® — Nalbuphine HCl 20mg, IM injection
  Other Names: Nalbuphine HCl
  Arms: Period I (reference drug)
Drug: SDE — Sebacoyl Dinalbuphine Ester 150mg/2ml, IM injection
  Other Names: Sebacoyl Dinalbuphine Ester Injection; LT1001
  Arms: Period II (Test drug)

SUMMARY:
This study is to evaluate the relative bioavailability of nalbuphine after single IM injection of Sebacoyl Dinalbuphine Ester (SDE) injection and Bain®, Nalbuphine HCl IM injection in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male or female adults in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
2. Vital signs (after 3 minutes resting in a upright position) which are within the following ranges:

   Ear body temperature between 35.0-37.5°C. Systolic blood pressure, 90-140 mm Hg. Diastolic blood pressure, 50-90 mm Hg. Pulse rate, 50-90 bpm. Fasting blood glucose, < 110 mg/dL.
3. Within -20% to +20% of the ideal body weight. For male subjects, body weight must be above 50 kg and for female subjects, body weight must be above 45 kg.
4. Able to sign informed consent prior to study.
5. Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

1. Use of any alcohol-containing products, prescription medications or over-the-counter, non-prescription preparations (including herbal preparations) within 2 weeks prior to study entry unless deemed acceptable by the Investigator (except up to 5 doses of ≤ 1000 mg of acetaminophen or ≤ 400 mg ibuprofen within this 2 week period).
2. Alcohol or caffeine ingested within 48 hours prior to dosing.
3. Significant illness within 2 weeks prior to dosing.
4. Participation in any clinical investigation within 2 months prior to dosing or longer as required by local regulation.
5. Donation or loss of more than 500 mL of blood within 3 months prior to dosing. Donation or loss of more than 250 mL of blood within 2 months prior to dosing.
6. Presence of cardiovascular disease.
7. Presence of gastrointestinal disease.
8. Presence of asthma or lung disease.
9. Presence of liver disease or liver injury as indicated by an abnormal liver function profile such as AST, ALT, gamma-GT, Alkaline Phosphatase, or Total Bilirubin. (value of AST or ALT above 3 times of the upper limit of the normal range; other items clinically significant abnormality judged by investigator).
10. Presence of impaired renal function as indicated by abnormal creatinine or BUN values or abnormal urinary constituents. (value of creatinine or BUN beyond the range from -20% of the lower limit of the normal range to +20% of the upper limit of the normal range; other items clinically significant abnormality judged by investigator)
11. Presence of neurological disease.
12. Presence of psychiatric disease.
13. Subject is positive for HIV immunology test.
14. A known hypersensitivity to nalbuphine or its analogs.
15. History of drug or alcohol abuse within 12 months prior to dosing.
16. Permanent confinement to an institution.
17. Pregnant or lactating women.
18. Individuals are judged by the investigator or pharmacokineticist to be undesirable as subjects for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Blood concentration of Nalbuphine HCl | Period I: pre-dose (0 h) and 0.083, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose for Bain®, Nalbuphine HCl IM injection ; Period II: pre-dose (0 h) and 6, 12, 24, 48, 72, 96, 120, 168, 216, 264 and 336 hours post dose for SDE IM injection
  Protocol-specified pharmacokinetic parameters will be determined from blood samples collected after each administration of study drug to assess the relative bioavailability of SDE.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, New Taipei City, Taiwan